CLINICAL TRIAL: NCT05682807
Title: Caffeine Versus Probiotic as Adjuvant Therapy for Preterm Neonates With Bronchopulmonary Dysplasia
Brief Title: Effect of Caffeine Versus Probiotic on Preterm Neonates With Bronchopulmonary Dysplasia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Ehab Fawzy Mohamed, clinical pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: caffeine probiotic BPD
Record Dates: First submitted 2022-10-14; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Caffeine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (group I) (No Intervention): will include 30 preterm neonates with BPD who will receive traditional therapy of BPD including minimizing exposure to oxygen, ventilation strategies, adequate nutrition and prudent administration of fluids
- caffeine group (group II) (Active Comparator): will include 30 preterm neonates with BPD who will receive traditional therapy of BPD in association with caffeine by intravenous route at a dose of 20 mg/kg loading dose with a 5-10 mg/kg/day maintenance dose given after 24 h ( Yuan et al., 2022) until discharge from the unit after clinical and laboratory improvement after two months.
  Interventions: Drug: Caffeine
- probiotic group (group III) (Active Comparator): will include 30 preterm neonates with BPD who will receive traditional therapy of BPD in association with probiotics sachets supplementation orally, in the form of lyophilized lactic acid bacteria each Aluminium stick pack contains 100 mg ( Meyer et al., 2020) Probio Tec BB12-Blend 30- IF* (SANDOZ®.) mixed with 10 ml sterile water and given by Ryle tube once daily until discharge from the unit after clinical and laboratory improvement after two months
  Interventions: Drug: Probiotic Formula

INTERVENTIONS:
Drug: Caffeine — 5-10 mg/kg/day IV maintenance dose given after 24 h for 2 months.
  Arms: caffeine group (group II)
Drug: Probiotic Formula — probiotics sachets supplementation orally, in the form of lyophilized lactic acid bacteria each Aluminium stick pack contains 100 mg ( Meyer et al., 2020) Probio Tec BB12-Blend 30- IF* (SANDOZ®.) mixed with 10 ml sterile water and given by Ryle tube once daily until discharge from the unit after clinical and laboratory improvement after two months.
  Arms: probiotic group (group III)

SUMMARY:
The aim of this study is to evaluate the effectiveness of caffeine versus probiotics supplementation as adjuvant therapy for preterm neonates with Bronchopulmonary dysplasia (BPD).

ELIGIBILITY:
Inclusion Criteria:

* Male and female preterm neonates less than 37 weeks gestational age.
* Suffering from Bronchopulmonary dysplasia (BPD) diagnosed as follow:
* History: Preterm infant with persistence oxygen dependency up to 28 days of life.
* Clinical signs: increase work of breathing, increase oxygen requirements , increase in apnea , bradycardia and retraction.
* Laboratory: arterial blood gases and electrolytes.
* Radiology: streaky interstitial markings, patchy atelectasis , intermingled with cystic areas and severe lung hyperinflation.

Exclusion Criteria:

* Term and post term neonates
* Neonates with congenital infections
* Neonates with major congenital anomalies

Ages: 0 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Complete blood count | 2 months
  Changes in blood parameters at baseline and after 2 months
Kidney function test | 2 months
  Changes in creatinine clearance at baseline and after 2 months
Liver function test | 2 months
  Changes in aspartate aminotransferase and alanine aminotransferase at baseline and after 2 months
Inflammatory parameter | 2 months
  changes in serum C-reactive protein at baseline and after 2 months

SECONDARY OUTCOMES:
change in Serum Tumor necrosis factor alpha (TNF-α) | 2 months
  blood sample will be collected at baseline and after 2 months
change in serum transforming growth factor (TGF)-β. | 2 months
  blood sample will be collected at baseline and after 2 months
change in Serum superoxide dismutase (SOD) | 2 months
  blood sample will be collected at baseline and after 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El Gharbia, Egypt